CLINICAL TRIAL: NCT02618057
Title: Effects of Oral Steroid in Mycoplasma Pneumoniae Pneumonia With Lobar Consolidation or Pleural Effusion in Children
Brief Title: Effects of Oral Steroid in Mycoplasma Pneumoniae Pneumonia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH_P01
Record Dates: First submitted 2015-11-08; First posted 2015-12-01 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Mycoplasma Pneumoniae Pneumonia
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Prednisolone; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid (Experimental): Prednisolone, 1.0 mg/kg/day, PO, for 5 days Levofloxacin, 10mg/kg/day, IV, for 5days
  Interventions: Drug: Prednisolone; Drug: Levofloxacin
- Control (Active Comparator): Levofloxacin, 10mg/kg/day, IV, for 5days
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Prednisolone — PO prednisolone, 1 mg/kg/day, for 5 days
  Other Names: Solondo
  Arms: Steroid
Drug: Levofloxacin — Levofloxacin, 10mg/kg/day, IV, for 5days

SUMMARY:
Mycoplasma pneumoniae is one of the most common causes of community-acquired pneumonia in children. The clinical course is typically self-limited and benign; however, rare cases of severe pneumonia can develop despite appropriate antibiotic therapy. The investigators aim to study the effects of prednisolone on severe M. pneumoniae pneumonia with lobar consolidation or pleural effusion in children.

DETAILED DESCRIPTION:
Mycoplasma pneumoniae is one of the most common causes of community-acquired pneumonia in children. The clinical course is typically self-limited and benign; however, rare cases of severe pneumonia can develop despite appropriate antibiotic therapy. The investigators aim to study the effects of prednisolone on severe M. pneumoniae pneumonia with lobar consolidation or pleural effusion in children. Participants will be randomly assigned (1:1 ratio) to receive either prednisone 1 mg/kg/d daily for 5 days or none. The primary endpoint was fever duration and analysed by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Mycoplasma pneumoniae infection
* Lobar pneumonia or pneumoniae with pleural effusion

Exclusion Criteria:

* Immunosuppresant host
* Chronic cardiovascular/pulmonary disease
* Hospital acquired infection

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fever duration | within the first 14 days after intervention

SECONDARY OUTCOMES:
Number of patients improved in chest X-ray | within the first 7 days after intervention
Number of patients with side effect of steroid | within the first 14 days after intervention
Number of patients improved in chest X-ray | within the first 14 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eun Hwa Choi, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea